CLINICAL TRIAL: NCT01424826
Title: A Single Arm, 3 Phase Study to Determine the Effect of Intermittent Dosing of Rifampicin on the Pharmacokinetics of Raltegravir in Healthy Volunteers
Brief Title: The Effect of Intermittent Rifampicin on Raltegravir
Acronym: RIFRAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helen Reynolds (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Helen Reynolds, Research Nurse, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoL000643; 2010-021461-73 (EudraCT Number)
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: HIV; Tuberculosis
Keywords: Healthy volunteers
MeSH Terms: conditions — Tuberculosis | interventions — Raltegravir Potassium; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Raltegravir — 400 mg bd for minimum of 28 days and maximum 35 days
Drug: Rifampicin — < 50 kg 600 mg 3 times/week for a minimum of 27 days and maximum of 34 days > 50 kg 900 mg 3 times/week for a minimum of 27 days and maximum of 34 days
Drug: Raltegravir — 800 mg bd for 4 days

SUMMARY:
This study seeks to address the question of whether intermittent dosing of rifampicin influences the pharmacokinetics of raltegravir when co-administered. This study aims to look at what happens when rifampicin is taken 3 times a week with the standard dose and an increased dose of raltegravir. This is to find out the best dose of raltegravir to take when taking rifampicin 3 times a week. The study will be conducted in 18 healthy volunteers.

DETAILED DESCRIPTION:
The aim of this study is to optimise the dosing of raltegravir when coadministered intermittently with rifampicin. The co-administration of rifampicin and antiretrovirals (ARVs) is both complicated and problematic due to the potent induction of metabolism by rifampicin. Rifampicin induces cytochrome P450 (CYP) enzymes, which results in reduced plasma concentrations of two groups of ARVs, the protease inhibitors (PIs) and the non-nucleoside reverse transcriptase inhibitors (NNRTIs). This pharmacokinetic interaction precludes the use of PIs and severely compromises the effectiveness of the NNRTI, nevirapine, as it potentially results in the loss of antiviral activity due to sub-therapeutic concentrations which will also lead to antiretroviral resistance.

Rifampicin also induces phase II enzymes including UDP-glucuronosyl transferase. The HIV integrase inhibitor, raltegravir, is primarily metabolised by UGT1A1 and therefore, there is the potential for a pharmacokinetic drug interaction with rifampicin. In fact, previous studies have shown a decrease in raltegravir AUC, CMAX, and C12 when co-administered with daily rifampicin. During directly observed therapy (DOTs) for TB, rifampicin is often given intermittently (e.g. 3 times a week). Although several studies have examined the interaction between raltegravir and daily rifampicin, currently there are no data regarding the pharmacokinetics of raltegravir when rifampicin is co-administered intermittently.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
* ≥ 18 years
* Male or female subjects
* A female may be eligible to enter and participate in the study if she:
* Is of non-child-bearing potential defined as ether post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age)or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or
* Is of child-bearing potential with a negative pregnancy test at screening and agrees to use one of the following methods of contraception to avoid pregnancy
* Complete abstinence from intercourse from 2 weeks prior to administration of IP, throughout the study and for at least 4 weeks after discontinuation of all study medication
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Any intrauterine device (IUD) with published data showing that the expected failure rate is < 1 % per year
* Any other method with published data showing that the expected failure rate is < 1 % PER YEAR
* Hormonal contraception plus a barrier method. Hormonal contraception alone will not be considered adequate for inclusion into or participation in this study due to one of the study drugs being rifampicin.

All subjects participating in the study will be counseled on safer sexual practices including the use of effective barrier methods (e.g. male condom)

Exclusion Criteria:

* Any significant acute or chronic medical condition
* Pregnant or lactating women
* Women of childbearing age unless using non hormonal contraception
* Males who are not using contraception
* Evidence of organ dysfunction or any clinically significant deviation from normal during screening including laboratory determinations such as abnormal LFTs
* Positive blood screen for HIV-1 and 2 antibodies
* Positive blood screen for hepatitis B or C antibodies
* Positive IGRA screen for TB
* Current or recent (within 3 months) gastrointestinal disease
* Clinically relevant alcohol or drug use or history of alcohol or drug use that will hinder compliance with treatment, follow up procedures or evaluation of adverse effects
* Use of proton pump inhibitors
* Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug
* Consumption of grapefruit and Seville oranges or products containing grapefruit or Seville oranges within 1 week of first study drug and for the duration of the study
* Use of any other drugs including over-the-counter medications and herbal preparations, within 2 weeks prior to first dose of study drug
* Previous allergy to any of the constituents of the pharmaceuticals in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in raltegravir area under the curve (AUC) 0-12h | Day 28 and day 33

SECONDARY OUTCOMES:
Number of participants with adverse events | 40 days (up to + 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Saye Khoo, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool & Broadgreen Univeristy Hospitals NHS Trust, Liverpool, United Kingdom

REFERENCES:
- [Derived] Reynolds HE, Chrdle A, Egan D, Chaponda M, Else L, Chiong J, Back DJ, Khoo SH. Effect of intermittent rifampicin on the pharmacokinetics and safety of raltegravir. J Antimicrob Chemother. 2015 Feb;70(2):550-4. doi: 10.1093/jac/dku376. Epub 2014 Sep 26. PMID 25261424